CLINICAL TRIAL: NCT01841346
Title: The First Jordanian Percutaneous Coronary Intervention (PCI) Registry
Brief Title: The First Jordanian PCI Registry: Events at 1 Year
Acronym: JoPCR1
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: JoPCR1-12-12-12
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Outcome after PCI; Middle Eastern Patients
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PCI patients: Patients undergoing PCI for elective or ACS will be enrolled.
  Interventions: Procedure: Procedure: PCI

INTERVENTIONS:
Procedure: Procedure: PCI
  Other Names: PCI (percutaneous coronary intervention)will be performed according to cardiologists discretion, with no randomization of stent types or medications.

SUMMARY:
The investigators will look at the short- (in hospital) and long- term ( 1 year)outcome in consecutive patients who undergo stent implantation and angioplasty in Jordan.

DETAILED DESCRIPTION:
1. Voluntary registry of consecutive patients undergoing Percutaneous coronary intervention (PCI).
2. Patients will be treated according to the treating cardiologists' discretion. No randomization of any medication or stent.
3. Baseline data on admission will be collected (cardiovascular risk factors, blood lipids, ect).
4. PCI procedure details and complications will be documented during the index admission.
5. Outcome events (death, MI, revascularization, stent thrombosis) will be evaluated at 1, 6, and 12 months by clinic visits or phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive PCI patients
* Arab nationality

Exclusion Criteria:

* less than 18 year of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute coronary syndrome and stable coronary syndromes undergoing PCI.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | 1 year
  All cases of deaths from cardiovascular causes will be counted at 1 year.

SECONDARY OUTCOMES:
Admission for urgent coronary revascularization | 1 year
  All events of hospital readmission for repeat coronary intervention for acute coronary syndrome from the time of discharge from hospital up to 1 year will be documented.

OTHER OUTCOMES:
Stent thrombosis | 1 year
  All cases of definite/probable/possible stent thrombosis will be documented from the time of stent implantation during the index admission to 1 year.
Baseline risk factors and outcome after 1 year | 1 year
  Several factors at baseline will be evaluated as potential contributors to adverse outcome after one year, including: age, gender, renal impairment, heart failure, CRUSADE bleeding risc score, GRACE risk score, diabetes, multiple risk factors, BMI, and smoking.
Adherence to guidelines in patients undergoing PCI | 1 year
  Using medications (statins, antiplatelets, ACI inhibitors/ARBs, B blockers, etc),and diagnostic and interventional procedures, and reaching target parameters (LDL cholesterol and HbA1c) according to the published guidelines will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari Hospital, Amman, Jordan

REFERENCES:
- See also: JCC group websites describes the studies done by the JCC Group — http://www.jcc-group.com